CLINICAL TRIAL: NCT03369210
Title: Liberal Transfusion Strategy to Prevent Mortality and Anaemia-associated, Ischaemic Events in Elderly Non-cardiac Surgical Patients
Brief Title: Liberal Transfusion Strategy in Elderly Patients
Acronym: LIBERAL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Patrick Meybohm, M.D., Prof. Dr. Patrick Meybohm, Wuerzburg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 139/17F
Record Dates: First submitted 2017-11-27; First posted 2017-12-11 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Transfusion-dependent Anemia; Surgery; Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liberal (Experimental): Liberal group (patients receive a RBC unit each time Hb falls ≤ 9 g/dl (≤ 5.6mmol/l) with a target range for the post-transfusion Hb level of 9-10.5 g/dl (5.6-6.5 mmol/l)).
  Interventions: Drug: red blood cell transfusion trigger
- Restrictive (Active Comparator): Restrictive group (patients receive a single RBC unit each time Hb falls ≤ 7.5 g/dl (≤ 4.7 mmol/l) with a target range for the post-transfusion Hb level of 7.5-9 g/dl (4.7-5.6 mmol/l).
  Interventions: Drug: red blood cell transfusion trigger

INTERVENTIONS:
Drug: red blood cell transfusion trigger — patients receive a RBC unit with different target ranges for the post-transfusion Hb levels

SUMMARY:
In this prospective, multicentre, open, randomised, controlled clinical trial elderly patients (≥ 70 years) undergoing intermediate- or high-risk non-cardiac surgery will be randomised either to a liberal group (patients receive a RBC unit each time Hb falls ≤ 9 g/dl (≤ 5.6mmol/l) with a target range for the post-transfusion Hb level of 9-10.5 g/dl (5.6-6.5 mmol/l)) or restrictive group (patients receive a single RBC unit each time Hb falls ≤ 7.5 g/dl (≤ 4.7 mmol/l) with a target range for the post-transfusion Hb level of 7.5-9 g/dl (4.7-5.6 mmol/l). Primary efficacy endpoint: is a composite of death from any cause and anaemia-associated, ischaemic events (defined as acute myocardial infarction, acute ischaemic stroke, acute kidney injury stage III, acute mesenteric ischaemia, acute peripheral vascular ischaemia) within 90 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 70 years of age scheduled for intermediate- or high-risk non-cardiac surgery will be registered
* Registered patients will be randomised only if they indeed develop severe anaemia (if Hb level falls ≤ 9 g/dl) during surgery (=day 0) or day 1, 2, or 3 after surgery

Exclusion Criteria:

* preoperative Hb level ≤ 9 g/dl
* chronic kidney disease requiring dialysis
* suspected lack of compliance with follow-up procedures
* participation in other interventional trials
* expected death within 3 months
* inability to provide informed consent with absence of a legally authorised representative/ legal guardian
* temporary inability to provide informed consent
* previous participation in our trial
* patients who are prevented from having blood and blood products according to a system of beliefs (e.g. Jehovah's Witnesses)
* preoperative autologous blood donation.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2470 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a composite endpoint | 90 days
  Composite of death and anaemia-associated events I. All-cause mortality defined as death from any cause. II. Acute myocardial infarction confirmed by a cardiologist III. Acute ischaemic stroke confirmed by a neurologist IV. Acute kidney injury (stage III) defined according to the Kidney Disease Improving Global Outcomes criteria: Increase of plasma creatinine level ≥ 3 times within a time window of 7 days or initiation of renal replacement therapy.
  V. Acute mesenteric ischaemia defined as ischaemia confirmed by intervention (abdominal surgery or mesenteric angiography).
  VI. Acute peripheral vascular ischaemia defined as a new non-thrombotic compromised circulation in a limb confirmed by angiography and/or leading to surgery.

SECONDARY OUTCOMES:
Proportion of patients receiving red blood cell transfusion | hospital discharge (an anticipated average of 10 days)
Number of red blood cell units transfused | hospital discharge (an anticipated average of 10 days)
Total length of stay in the intensive care unit | hospital discharge (an anticipated average of 10 days)
Total length of stay in hospital | hospital discharge (an anticipated average of 10 days)
Number of participants with acute kidney injury stage I-II | hospital discharge (an anticipated average of 10 days)
  The occurrence of acute kidney injury (stage I or II) defined according to the Kidney Disease Improving Global Outcomes criteria (stage I: increase of plasma creatinine level ≥ 1.5-1.9 times baseline or ≥ 0.3mg/dl within 48 hours; stage II: increase of plasma creatinine level ≥ 2-2.9 times baseline within a time window of 7 days) during the initial hospital stay
Time to infection | 90 days
  Time to (first) infection (infection requiring therapeutic intravenous antibiotic treatment (pneumonia, wound infection, sepsis, central line associated blood stream infection)) during the initial hospital stay or leading to hospital re-admission
Time to re-hospitalisation | 90 days
  Time to (first) re-hospitalisation
functional status (Barthel index) | 90 days
  Functional status (assessed by Barthel Index)
Health-related quality of life | 90 days
  Health-related quality of life (assessed by EuroQoL EQ-5D and 12-item World Health Organisation Disability Assessment Schedule WHODAS 2.043) by telephone questionnaire)
Occurrence of any individual component of the composite | 1 year
  composite components (all-cause mortality, acute myocardial infarction, acute stroke, acute kidney injury stage III, acute mesenteric ischaemia, and/or acute peripheral vascular ischaemia)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Meybohm, MD, Principal Investigator — Wuerzburg University Hospital
Locations (14):
- Germany (14):
  - University Hospital Augsburg, Augsburg
  - Berlin Charite CCM, Berlin
  - Charite Berlin CBF, Berlin
  - University Hospital Bonn, Bonn
  - Klinikum Dortmund, Dortmund
  - University Hospital Frankfurt, Frankfurt
  - University Hospital Hamburg, Hamburg
  - University Hospital Jena, Jena
  - University Hospital Schleswig-Holstein, Kiel
  - University Hospital Mainz, Mainz
  - St. Franziskus Hospital Münster, Münster
  - University Hospital Münster, Münster
  - University Hospital Regensburg, Regensburg
  - University Hospital Würzburg, Würzburg

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Meybohm P, Lindau S, Treskatsch S, Francis R, Spies C, Velten M, Wittmann M, Gueresir E, Stoppe C, Kowark A, Coburn M, Selleng S, Baschin M, Jenichen G, Meersch M, Ermert T, Zarbock A, Kranke P, Kredel M, Helf A, Laufenberg-Feldmann R, Ferner M, Wittenmeier E, Gurtler KH, Kienbaum P, de Abreu MG, Sander M, Bauer M, Seyfried T, Gruenewald M, Choorapoikayil S, Mueller MM, Seifried E, Brosteanu O, Bogatsch H, Hasenclever D, Zacharowski K; LIBERAL Collaboration Group. Liberal transfusion strategy to prevent mortality and anaemia-associated, ischaemic events in elderly non-cardiac surgical patients - the study design of the LIBERAL-Trial. Trials. 2019 Feb 4;20(1):101. doi: 10.1186/s13063-019-3200-3. PMID 30717805
- See also: Related Info — http://www.liberal-trial.de